CLINICAL TRIAL: NCT04919603
Title: Impact of Exercise Intervention on the Phenome (Metabolism and Predictive Complications) in Well Characterised Pre-diabetes and New Onset Type 2 Diabetes Cohorts in China
Brief Title: Impact of Exercise Intervention on the Phenome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.0/2020-07-29
Record Dates: First submitted 2021-04-22; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Overweight and Obesity; Physical Activity
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced physical activity group (Experimental): the participants will take high-intensity exercise in accordance with High Intensity Interval Training (HIIT) prescriptions, with maximum heart rate and relative maximal oxygen uptake monitored. They will take both aerobic and resistance training exercise consecutively, and total training time will be expected to reach at least 150 minutes per week.
  Interventions: Behavioral: Enhanced physical activity intervention
- Standard education group (Experimental): the participants will receive no extra intervention but diabetes health education, which will be carried out in large classrooms, in groups, and over the telephone. The education is mainly consisted of instructions on diabetes prevention according to < Guidelines for prevention and treatment of type 2 diabetes in China (2017 edition)telephone. The education is mainly consisted of instructions on diabetes prevention according to < Guidelines for prevention and treatment of type 2 diabetes in China (2017 edition)>.
  Interventions: Behavioral: Standard education

INTERVENTIONS:
Behavioral: Enhanced physical activity intervention — the participants will take high-intensity exercise in accordance with High Intensity Interval Training (HIIT) prescriptions, with maximum heart rate and relative maximal oxygen uptake monitored. They will take both aerobic and resistance training exercise consecutively, and total training time will be expected to reach at least 150 minutes per week.
  Arms: Enhanced physical activity group
Behavioral: Standard education — the participants will receive no extra intervention but diabetes health education, which will be carried out in large classrooms, in groups, and over the telephone. The education is mainly consisted of instructions on diabetes prevention according to < Guidelines for prevention and treatment of type 2 diabetes in China (2017 edition)
  Arms: Standard education group

SUMMARY:
It is an open-label, parallel-group, randomized controlled clinical trial, which is designed to enroll people with different glucose metabolism status who are also overweight or obese, including people with normal glucose metabolism, pre-diabetes patients and newly diagnosed type 2 diabetes patients. The patients are randomized to an enhanced physical activity intervention (high-intensity interval training exercise prescription combined with resistance training) or standard education group (diabetes health education only, including lifestyle education and guidance) for 12 weeks. This trial intends to compare the influence of enhanced physical activity treatment with that of a standard education on liver steatosis, serum glucose and lipids level, insulin sensitivity, cardiovascular metabolic parameters, metabolic molecules, and gut microbiota profile et al.

DETAILED DESCRIPTION:
The trial will recruit 270 patients from 2 hospitals within the China Diabetes Clinical Research Network. Eligible criteria include men and women aged 18-65 years; with normal glucose metabolism or pre-diabetes or newly diagnosed type 2 diabetes; no insulin treatment; BMI ≥23 kg/m2 and <40 kg/m2. Main exclusion criteria include severe cardiovascular diseases, uncontrolled hypertension, and other serious illness. The proposed trial has 90% statistical power to detect an absolute 3.0% reduction of liver triglyceride level changes between intensive physical activity intervention and standard education groups at a 2-sided significance level of 0.05. To achieve the proposed study objectives, we plan to perform the following specific aims:

1. Recruit 270 study participants who meet the eligibility criteria, including 90 people with normal glucose metabolism, 90 pre-diabetes patients and 90 newly diagnosed type 2 diabetes patients, and randomly assign 135 to the enhanced physical activity intervention group and 135 to the standard education group for 12 weeks;
2. Employ a study-wide strategy to encourage standard of care for all participants for the treatment of type 2 diabetes and other metabolic disorders;
3. Obtain clinical data on study outcomes for up to 12 months of follow-up among all trial participants;
4. Perform strict quality control procedures for intervention and data collection;
5. Conduct data analysis according to the intention-to-treat principle;
6. Disseminate the study findings to influence clinical practice and clinical guidelines.

The results will be analyzed to examine the pan-omics changes after the interventions and clarify their predictive benefits on the effects of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-65 years;
2. Normal glucose metabolism or pre-diabetes or newly diagnosed type 2 diabetes

   Normal glucose metabolism:
   * FBG<5.6mmol/L and
   * 2h-PG<7.8mmol/L and
   * HbA1c<5.7%;

   Pre-diabetes:
   * 5.6mmol/L ≤ FBG ≤ 6.9mmol/L and/or
   * 7.8mmol/L ≤ 2h-PG ≤ 11.0mmol/L and/or
   * 5.7% ≤ HbA1c ≤ 6.4%;

   Newly diagnosed diabetes:

   o Duration of type 2 diabetes is less than 5 years;
3. No insulin treatment;
4. 23 Kg/m2 ≤ Body mass index (BMI) <40 Kg/m2;

Exclusion Criteria:

Eligibility Minimum Age: 18 Years Maximum Age: 65 Years Sex: All Gender Based: No Accepts Healthy Volunteers: No

Criteria: Inclusion Criteria:

1. Men and women aged 18-65 years;
2. Normal glucose metabolism or pre-diabetes or newly diagnosed type 2 diabetes

   Normal glucose metabolism:
   * FBG<5.6mmol/L and
   * 2h-PG<7.8mmol/L and
   * HbA1c<5.7%;

   Pre-diabetes:
   * 5.6mmol/L ≤ FBG ≤ 6.9mmol/L and/or
   * 7.8mmol/L ≤ 2h-PG ≤ 11.0mmol/L and/or
   * 5.7% ≤ HbA1c ≤ 6.4%;

   Newly diagnosed diabetes:

   o Duration of type 2 diabetes is less than 5 years;
3. No insulin treatment;
4. 23 Kg/m2 ≤ Body mass index (BMI) <40 Kg/m2;

Exclusion Criteria:

1. Severe cardiovascular disease:

   * current angina
   * myocardial infarction or stroke within last six months
   * heart failure (NYHA grading III~IV)
   * symptomatic periphery vascular disease
2. Uncontrolled hypertension: systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg;
3. Myocardial ischemia indicated by resting ECG;
4. Cardiac dysfunction indicated by Echocardiogram;
5. Abnormal HS-TNT or NT-proBNP concentration;
6. Foot ulcers, peripheral neuropathy or skeletal disorders;
7. Taking high intensity exercise more than 75 minutes or moderate intensity exercise more than 150 minutes per week during the screening phase
8. ALT or AST levels more than three times the upper limit of the normal range or active liver diseases;
9. eGFR <60 ml/min/1.73 m2, or serum creatinine >1.5 mg/dl for men or 1.3mg/dl for women; or macro albuminuria (urine albumin/creatinine>300mg/g)
10. Malignant tumor in active-stage, or in remission stage but less than 5 years from the most recent treatment
11. Past or present confirmed psychiatric illness or drug dependence;
12. Currently taking medications known to affect weight (e.g. anti thyroid drugs, glucocorticoids);
13. Known to have weight-affecting diseases (e.g. malabsorption, functional bowel disease, uncontrolled low sodium/hyperthyroidism, eating disorders);
14. Known to have metabolism-affecting diseases;
15. Other acute diseases supported by clinical evidence which may contradict to the interventions;
16. Pregnancy, currently trying to become pregnant, or of child-bearing potential and not using birth control;
17. Currently participating in another intervention study;
18. Failure to obtain informed consent from participant;
19. Any factors judged by the clinic team to be likely to limit adherence to interventions;
20. Any other medical condition judged by the clinic team not eligible for the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in liver steatosis quantified by MRI-PDFF (percentage) | 12 weeks

SECONDARY OUTCOMES:
Change in liver steatosis quantified by MRI-PDFF (percentage) | 1 year
Change in the level of fasting blood glucose (mmol/l) | 12 weeks and 1 year
Change in the level of plasma glucose of 2 hours post glucose-load (mmol/l) | 12 weeks and 1 year
Change in the level of HbA1c (percentage) | 12 weeks and 1 year
Change in body mass index (BMI) | 12 weeks and 1 year
  Body weight (kg) and height (m) will be combined to report BMI in kg/m^2
Change in waist circumstance (cm) | 12 weeks and 1 year
Change in body fat level (%) | 12 weeks and 1 year
  Quantified by bioelectrical impedance analysis in a human body composition analyzer
Change in serum non-HDL-C level (mg/dl) | 12 weeks and 1 year
Change in serum total cholesterol level (mg/dl) | 12 weeks and 1 year
Change in serum VLDL-C level (mg/dl) | 12 weeks and 1 year
Change in serum LDL-C level (mg/dl) | 12 weeks and 1 year
Change in serum HDL-C level (mg/dl) | 12 weeks and 1 year
Change in serum ApoB level (mg/dl) | 12 weeks and 1 year
Change in basal metabolic rate (BMR) (Kcal) | 12 weeks and 1 year
  Quantified by bioelectrical impedance analysis in a human body composition analyzer
Change in blood pressure (mmHg) | 12 weeks and 1 year
Change in heart rate | 12 weeks and 1 year
Change in insulin sensitivity | 12 weeks and 1 year
  Quantify by HOMA score, which is calculated multiplying fasting plasma insulin (FPI, mIU/L) by fasting plasma glucose (FPG, mmol/L), then dividing by the constant 22.5, i.e. HOMA-IR = (FPI×FPG)/22.5.
Change in islet β-cell function | 12 weeks and 1 year
  Quantify by HOMA score, which is calculated with fasting plasma insulin (FPI, mIU/L) and fasting plasma glucose (FPG, mmol/L), i.e. HOMA-β = 20*FPI/(FPG-3.5).
Change in serum fetuin-A concentration (μg/mL) | 12 weeks and 1 year
Change in serum GREM2 concentration (pg/ml) | 12 weeks and 1 year
Change in gut hormones, monocyte subtypes and other serum biomarkers | 12 weeks and 1 year
Change in metabolic molecules concentration | 12 weeks and 1 year
Change in microRNA concentration | 12 weeks and 1 year
Change in overall gut microbiota profile | 12 weeks and 1 year
  change in gut microbiota composition and proportion of specific gut flora.
Depression | 12 weeks and 1 year
  Evaluated with PHQ-9 scores. The PHQ is 59-question instrument, referring to the level of interest in doing things, feeling down or depressed, difficulty with sleeping, energy levels, eating habits, self-perception, ability to concentrate, speed of functioning and thoughts of suicide. Responses range from "0" (Not at all) to "3" (nearly every day).The total sum of the responses suggests varying levels of depression. Scores range from 0 to 27. In general, a total of 10 or above is suggestive of the presence of depression.
Health related quality of life | 12 weeks and 1 year
  Evaluated with HQoL scales such as Short Form 12 Health Survey Questionnaire. The SF-12 is 12-question instrument, covering the eight domains of health outcomes, including physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 48. A higher score indicates a better health state.
Change in diet pattern | 12 weeks and 1 year
  Evaluated with a semiquantitative food frequency questionnaire.
Change in sleeping pattern | 12 weeks and 1 year
  Evaluated with Pittsburgh Sleep Quality Index, PSQI. Scores range from 0 to 21. A higher score indicates a worse sleeping pattern.
Change in daily exercise | 12 weeks and 1 year
  Evaluated with short form International Physical Activity Questionnaire (IPAQ).
Cardiovascular risk | 12 weeks and 1 year
  Evaluated with Framingham Risk Scores. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Institute of Endocrine and Metabolic Diseases, Shanghai, Shanghai Municipality
  - The Third People's Hospital of Datong City, Datong, Shanxi